CLINICAL TRIAL: NCT02882087
Title: A Phase II, Placebo-Controlled, Multicenter, Dynamic Randomized, Double Blind Trial of RC18, a Recombinant Human B Lymphocyte Stimulating Factor Receptor-Antibody Fusion Protein in Subjects With Inadequate Response of TNF-α Antagonists Due to Treat Moderate and Severe Rheumatoid Arthritis
Brief Title: A Study of the Efficacy and Safety of TACI-antibody Fusion Protein Injection (RC18) in Subjects With Inadequate Response to TNF-α Antagonists Due to Treat Moderate and Severe Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of trial population, unable to recruit subjects
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C004 RACLLI
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Moderate and Severe Rheumatoid Arthritis
MeSH Terms: conditions — Lymphoma, Follicular; Arthritis, Rheumatoid | interventions — Methotrexate; RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Comparator (Experimental): Placebo SC plus MTX. Patients received placebo SC weekly administered subcutaneously for 24 times.All patients had a foundation MTX therapy, MTX dose should be stable, not to adjust the dose.The researchers evaluated the efficacy of the patient in 12 week.Evaluation of efficacy in patients if not get the ACR20 response, adjust the treatment plan given the test drug.Test group continue to the test drug,placebo group switch to the test drug.
  Interventions: Drug: Placebo plus MTX
- Experimental: RC18 160 mg plus MTX (Experimental): Patients received the test group RC18 160mg weekly administered subcutaneously for 24 times. All patients had a foundation MTX therapy, MTX dose should be stable, not to adjust the dose.
  Interventions: Drug: RC18 160 mg plus MTX

INTERVENTIONS:
Drug: Placebo plus MTX — All patients had a foundation MTX therapy.The researchers evaluated the efficacy of the patient in 12 week.study investigator evaluate the patients of curative effect . The researchers evaluated the efficacy of the patient in 12 week.Evaluation of efficacy in patients if not get the ACR20 response, adjust the treatment plan given the test drug.Test group continue to the test drug,placebo group switch to the test drug.
  Other Names: MTX=Methotrexate
  Arms: Placebo Comparator
Drug: RC18 160 mg plus MTX
  Other Names: RC18; MTX=Methotrexate
  Arms: Experimental: RC18 160 mg plus MTX

SUMMARY:
This is a phase Ⅱ, placebo-controlled, multicenter, dynamic randomized, double blind study of the efficacy and safety of RC18, a recombinant human B lymphocyte stimulating factor receptor-antibody fusion protein in subjects with inadequate response of TNF-α antagonists due to treat moderate and severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult onset RA by a physician as defined by the 1987 and/or 2010 ACR criteria.and ESR or C - reaction protein ( CRP ) is greater than the normal range
* Aged 18-65 years old;
* Consent to use effective contraception during the study period (women of childbearing age)
* Patients with an inadequate response to existing therapies at least one anti-TNFs Infliximab (Remicade ) at least three times, adalimumab (Humira), at least four times, etanercept ( Enbrel) use at least 8 weeks, etanercept use at least 8 weeks .And Last medication time to randomization more than 12 weeks .
* Voluntarily signed informed consent ;
* Patients have been taking MTX for at least 12 weeks at the screening and maintaining dose stability ≥7.5mg/ weeks (or equivalent dose) 4weeks before randomization .
* If the subjects are taking DMARDs (except MTX) at screening, the test was discontinued for at least 4 weeks before randomization.
* If subjects are receiving treatment of corticosteroid ,must stabilize dose (dose of prednisone) at least equal to or less than 10mg / day for 4 weeks (before randomization);
* If subjects are receiving treatment of NSAIDs ,must stabilize dose (dose of prednisone) at least 4 weeks (before randomization).
* When the patient's condition to achieve moderate to severe active RA at the screening , defined as at least 6/68 tenderness joints and at least 6/66 swollen joints.

Exclusion Criteria:

-There are serious heart, liver, kidney and other important organs and blood, endocrine system diseases and medical history;

Evaluation criteria for severity :

1. liver function ≥2 ULN;
2. Cr >135μmol/L;
3. WBCs<3x 109/L;;
4. hemoglobin<85g/L;
5. platelet count<80x 109/L.

   * Have a historically active hepatitis or active hepatitis or medical history;HBsAg- surface antigen positive patients are not allowed to be selected, but only anti HBC single positive is added to do HBV-DNA quantitative detection, if the HBV-DNA quantity is negative can not be regarded as the exclusion;
   * Immune deficiency, uncontrolled severe infection and patients with active or recurrent peptic ulcer;
   * pregnant , lactating women and men or women who have birth plans in the past 6 months ;
   * Have a history of allergic reaction to contrast agent for parenteral administration and human biological medicines.
   * Receipt of live vaccine within 1 month(excepting for herpes zoster vaccine)
   * Have participated in any clinical trial in the first 28 days of the initial screening or 5 times half-life period of the study compound (taking the time for the elderly).
   * Patients with using of biological agents for the treatment of DMARDs within three months
   * Infection with herpes zoster or HIV virus at the screening;
   * Active TB at screening.Exception for patients with PPD≥15mm.But Patients with anti tuberculosis treatment for 3 years without relapse are allowed to participate in the trial;
   * Malignant tumor patients :the patients who suffering from malignant tumor has been removed and no recurrence or who with cervical carcinoma in situ have evidence of metastatic disease and with basal cell or squamous cell carcinoma had been completely removed and at least 3 years without recurrence can participate in .
   * there was a history of long-term alcohol abuse, intravenous drug abuse or other illicit drug abuse within 6 months
   * Planning to have surgery for RA or other significant surgery during the period of the study.
   * patients experienced any of the following events within 12 weeks before screening : myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association class IV heart failure
   * Patients received interferon treatment (such as interferon alpha, intron alpha, peg-intron, double talon, intergen, Pegasys etc.) within 4 weeks before screening , or are expected to test period will need to accept interferon therapy.
   * The combined use of immunosuppressive agents associated with organ transplantation is not allowed during the study period.
   * Combined with non RA any other systemic inflammatory diseases, including but not limiting to, juvenile chronic arthritis, vertebral arthrosis, limited enteritis (Crohn's disease), ulcerative colitis, psoriatic arthritis, activity of vasculitis or gout. But with secondary drying syndrome of patients need not be excluded.
   * Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each group reached ACR20 24 weeks for visits | Week 24（Visit 9 ）
  ACR20 response: Patients with tenderness and swollen joint counts and 20% improvement,At least 3 20% improvement in the following 5:a.Health Assessment Questionnaire;b.Subjects assessed pain VAS score;c.Assess the overall situation of the disease subject VAS score;d.Researchers assessed the overall situation of the disease in the VAS score;e.Acute phase reactants(ESR or CRP)

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Clinically Meaningful Improvement in Disease Activity Score 28 (DAS28)at week 12 and week 24. | week 12 and week 24
  DAS28 was calculated from the tender joint count (TJC) of 28 joints, swollen joint count (SJC) of 28 joints, erythrocyte sedimentation rate (ESR) (in millimeters [mm]/hour), and the participant's global assessment of disease activity (100 mm visual analog scale [VAS]: 0 mm=no disease activity to 100 mm=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56*square root (√) of TJC + 0.28*√(SJC) + 0.70*log natural (ESR) + 0.014*global assessment of disease activity (100 mm VAS). The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.

OTHER OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology ACR50 and ACR70 Responses at week 12 or week 24. | week 12 and week 24
Sharp score relative change from baseline at week 24 | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided